CLINICAL TRIAL: NCT05077995
Title: Validity and Reliability of the Polar M200 Activity Monitor to Measure Sedentary and Active Time
Brief Title: Validity and Reliability of the Polar M200 Activity Monitor
Acronym: VAPO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Responsible Party: Principal Investigator, Bert Op't Eijnde, Prof. dr., Hasselt University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: VAPO-UH
Record Dates: First submitted 2021-10-01; First posted 2021-10-14 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Healthy Persons; Fitness Trackers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy adult group (Experimental): Sixty healthy adults, aged 18-65 years, will be included following written informed consent.
  Interventions: Device: Polar M200

INTERVENTIONS:
Device: Polar M200 — Participants will have to wear the activity monitors (AP and Polar M200) for at least 7 days. Minutes spent in each activity type will be summed to a total day score. Participants will be instructed to do their regular daily life activities without limitation, but to note their main activity categories in an activity diary, with a main focus on cycling and participation in structured exercise.

SUMMARY:
The aim of this study will be to investigate the validity of a consumer available activity tracker (Polar M200) in free-living conditions to measure sedentary time.

DETAILED DESCRIPTION:
The aim of the present study is to evaluate the validity from a commercially available wearable Polar device. Consumer-based activity trackers are generally cheaper, designed for long-term wear and are less intrusive. Potentially, consumer-based activity trackers can be used for research purposes, but high-quality validation studies are needed. The aims of this study will be to assess validity of sedentary outcome measures of a Polar device during free-living conditions in comparison with the ActivPAL3TM activity monitor (AP; PAL Technologies Ltd, Glasgow, UK), which is considered the gold standard to measure sedentary time in free-living conditions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults

Exclusion Criteria:

* /

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-07-25 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Sedentary time | 7 days
  Sedentary time

SECONDARY OUTCOMES:
Steps | 7 days
  Number of steps
Sleeping time | 7 days
  Sleeping time
Standing time | 7 days
  Standing time
Walking time | 7 days
  Walking and running time

CONTACTS AND LOCATIONS:
Overall Officials: Bert Op 't Eijnde, Prof. dr., Principal Investigator — Hasselt University
Locations (1):
- Hasselt University, Hasselt, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: No